CLINICAL TRIAL: NCT03512392
Title: Role of Active Deresuscitation After Resuscitation- 2: a Pilot Randomised Controlled Trial of Conservative Fluid Management Versus Usual Care in Critical Illness
Brief Title: Role of Active Deresuscitation After Resuscitation-2
Acronym: RADAR-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17057JS-AS
Record Dates: First submitted 2017-12-05; First posted 2018-04-30 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Critical Illness; Sepsis; Trauma
Keywords: fluid therapy; furosemide; diuretics; Injections, Intravenous; Infusions, Intravenous; Spironolactone; Indapamide
MeSH Terms: conditions — Critical Illness; Sepsis; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Randomised, open-label, allocation concealed, pilot trial
Masking Description: Group assignment and early (up to 28 day) data will be locked and unavailable to investigators undertaking 6-month follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative fluid and deresuscitation (Experimental): * Fluid restriction (avoidance of maintenance intravenous fluid and minimisation of drug diluent volumes)
  * Daily assessment of eligibility for deresuscitation for 3 days (eligible if oedema in more than 1 site and cumulative fluid balance > 2 litres)
  * Deresuscitation to target negative daily fluid balance of 1 to 3 litres:
    5mg Indapamide daily (enteral) 100mg Spironolactone daily (enteral) 0.5mg/kg furosemide once (intravenous, max 40mg) 2.5-20mg/hr furosemide infusion titrated to effect OR continuous renal replacement therapy with fluid removal
  Interventions: Other: Conservative fluid and deresuscitation strategy
- Usual care (Active Comparator): Usual care at the discretion of the treating team
  Interventions: Other: Usual care strategy

INTERVENTIONS:
Other: Conservative fluid and deresuscitation strategy — Conservative administration of intravenous fluid and active deresuscitation using diuretics or renal replacement therapy for eligible patients
  Arms: Conservative fluid and deresuscitation
Other: Usual care strategy — Usual care at the discretion of the clinical team
  Arms: Usual care

SUMMARY:
RADAR-2 will be a randomised, open-label, allocation concealed, pilot trial of conservative fluid administration and deresuscitation compared with usual care in patients who are critically ill.

DETAILED DESCRIPTION:
The optimal approach to fluid balance in critically ill patients is uncertain. A recent systematic review found low quality evidence in favour of a conservative fluid or deresuscitative approach (active removal of accumulated fluid using diuretics and/or renal replacement therapy) compared with a liberal strategy or usual care. The RADAR-2 pilot randomised trial will compare conservative fluid and deresuscitation with usual care in patients who are mechanically ventilated in an intensive care unit. The main hypothesis is that in critically ill patients, a post-resuscitation fluid strategy comprising conservative fluid administration and active deresuscitation reduces net fluid balance, is safe and improves clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Invasive mechanical ventilation
2. Treating ICU doctor expects patient to require treatment in an ICU beyond the next calendar day
3. Between 24 and 48 hours from ICU admission at the time of randomisation

Exclusion Criteria:

1. Age < 16 years
2. Body weight <40kg (measured or estimated)
3. Diabetic ketoacidosis or Hyperosmolar hyperglycaemic state
4. Non-traumatic subarachnoid haemorrhage
5. Acute cardiac failure or cardiogenic shock
6. End-stage renal failure (on dialysis)
7. Known to be pregnant
8. Suspected or proven active diabetes insipidus (DDAVP within 24 hours)
9. Not expected to survive for 72 hours
10. Active 'Do not attempt resuscitation' order
11. Refusal of consent
12. Inability of personal consultee to understand written or verbal information and for whom no interpreter is available
13. Known allergy to one or more of the study drugs
14. Inability to measure fluid balance

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Day 3 fluid balance | From beginning of day 2 to the beginning of study day 3.
  Change in fluid balance (mL) between the beginning of study day 2 and the beginning of study day 3.

SECONDARY OUTCOMES:
Cumulative fluid balance | Up to the beginning of days 3 and 5, and at ICU discharge (estimated median day 7)
  Cumulative fluid balance (mL) from ICU admission
Incidence of significant protocol violations | Up to study day 5
  Incidence of significant protocol violations (total number of patients, per site, and by nature of protocol violation) up to day 5 (intervention period)
Incidence of reported adverse events | Up to study day 5
  Incidence of reported adverse events up to day 5 (intervention period)
Change in Sequential Organ Function Assessment scores | From baseline until day 3 and day 5
  Change in Sequential Organ Function Assessment scores from baseline, overall (0-24) and 6 individual organ sub scores (respiratory, cardiovascular, neurological, coagulation, renal and liver, each scored 0-4 which are added to give a total score). Higher values represent more deranged physiology and predict mortality for critically ill patients.
Mortality | 28 and 180 days
  Mortality
Duration of mechanical ventilation | 28 days
  Duration of mechanical ventilation in survivors and non-survivors (number of days or part thereof from initiation of mechanical ventilatory support until unassisted breathing)
Length of ICU stay | 28 days
  Length of ICU stay (number of days or part thereof from admission to an ICU or being under the care of a critical care team or consultant until ICU discharge)
Acute kidney injury | Up to day 5.
  Incidence of new acute kidney injury defined as estimated KDIGO Stage 3 (before and after correction for fluid balance)
Cognitive function | 180 days
  Cognitive function score (assessed using the Montreal Cognitive Assessment (MoCA-blind) instrument)
Health-related quality of life | 180 days
  Health-related quality of life (HR-QoL) (assessed using absolute values of a telephone-administered EQ-5D (EuroQoL 5 Dimension Scale) questionnaire). This has 5 domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, each of which are scored 1-5, with 1 being best and 5 being worst health. Each domain is reported separately. A total score is generated and is indexed to population reference values for that country (in this case UK) according to the time of data collection. It is therefore not possible to pre-specify a range for the indexed score.

OTHER OUTCOMES:
Mean regional cerebral oxygen saturation | 72 hours from randomisation
  Near infra-red spectroscopic measurement of regional cerebral oxygen saturation), mean rScO2 level (%)
Minimum regional cerebral oxygen saturation | 72 hours from randomisation
  Near infra-red spectroscopic measurement of regional cerebral oxygen saturation), Minimum rScO2 level
Regional cerebral hypoxia burden | 72 hours from randomisation
  Near infra-red spectroscopic measurement of regional cerebral oxygen saturation), proportion of time spent with rScO2 below thresholds of 50%, 65%, and 75% as a proportion of the time for which cerebral oxygenation is measured, expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Silversides, MB BCh, Principal Investigator — Belfast Health and Social Care Trust
Locations (8):
- United Kingdom (8):
  - Aneurin Bevan University Health Board, Newport, Gwent
  - Northern Health and Social Care Trust, Antrim, Northern Ireland
  - Belfast City Hospital, Belfast, Northern Ireland
  - Royal Victoria Hospital, Belfast, Northern Ireland
  - South-Eastern Health and Social Care Trust, Dundonald, Northern Ireland
  - Sunderland Royal Hospital, Sunderland, Tyne and Wear
  - Western Health and Social Care Trust, Londonderry
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silversides JA, Major E, Ferguson AJ, Mann EE, McAuley DF, Marshall JC, Blackwood B, Fan E. Conservative fluid management or deresuscitation for patients with sepsis or acute respiratory distress syndrome following the resuscitation phase of critical illness: a systematic review and meta-analysis. Intensive Care Med. 2017 Feb;43(2):155-170. doi: 10.1007/s00134-016-4573-3. Epub 2016 Oct 12. PMID 27734109
- [Result] Silversides JA, McMullan R, Emerson LM, Bradbury I, Bannard-Smith J, Szakmany T, Trinder J, Rostron AJ, Johnston P, Ferguson AJ, Boyle AJ, Blackwood B, Marshall JC, McAuley DF. Feasibility of conservative fluid administration and deresuscitation compared with usual care in critical illness: the Role of Active Deresuscitation After Resuscitation-2 (RADAR-2) randomised clinical trial. Intensive Care Med. 2022 Feb;48(2):190-200. doi: 10.1007/s00134-021-06596-8. Epub 2021 Dec 16. PMID 34913089

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/92/NCT03512392/SAP_001.pdf